CLINICAL TRIAL: NCT01687452
Title: Microparticles, Vector of Genetic Information During HIV Infection ?
Brief Title: Microparticles, Vector of Genetic Information During HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A00015-36; 2010-25 (Other: AP HM)
Record Dates: First submitted 2011-03-31; First posted 2012-09-19 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: HIV,
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Groupe A (Experimental): Infected by the HIV Innocents of antiretroviral treatment, with a viral plasmatique load > 1000 copies / ml
  Interventions: Biological: Blood samples
- group B (Experimental): Infected by the HIV whith antiretroviral treatment for at least 6 months,, with a viral plasmatique load > 40 copies / ml
  Interventions: Biological: Blood samples
- group C (Placebo Comparator): Healthy volunteers
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples

SUMMARY:
The aim of the investigators study is to demonstrate in healthy subjects and a cohort of patients infected with HIV, the presence of miRNAs in circulating peripheral blood microparticles (MPs).

ELIGIBILITY:
Inclusion Criteria:

* Age of 40 +/-10 years
* Seronegativity for the HIV 2
* Patients of the group A: seropositivity for the HIV 1 confirmed in ELISA and Western Blot for at least 2 years and having never received from antiretroviral treatment, with a viral plasmatique load > 1000 copies / ml
* Patients of the group B: seropositivity for the HIV 1 confirmed in ELISA and Western Blot for at least 2 years and under stable antiretroviral treatment for at least 6 months, with a viral load undetectable plasmatique (< 40 copies / ml)
* patients of the group C : Matching on the age (+/-3 years) to a patient
* Be considered healthy by the Investigator after a clinical examination Seronegativity for the HIV 1 confirmed in ELISA the day of the taking

Exclusion Criteria:

group A et B

* Age of < 30 years and > in 50 years
* Seropositivity for the HIV 2

group C Seropositivity for the HIV 2

- Be under medicinal treatment

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
NUMBER OF miRNAs | 2 YEARS

SECONDARY OUTCOMES:
Demonstrate the presence of miRNAs in microparticles | 2 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France